CLINICAL TRIAL: NCT00515099
Title: Effect of Antithymocyte Globulin on Preserving Beta Cell Function in New Onset Type 1 Diabetes Mellitus
Brief Title: Study of Antithymocyte Globulin for Treatment of New-onset T1DM
Acronym: START
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAIT ITN028AI
Record Dates: First submitted 2007-08-10; First posted 2007-08-13 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-04

CONDITIONS: New-onset Type 1 Diabetes Mellitus
Keywords: New-onset Type 1 Diabetes Mellitus; New-onset T1DM; New-onset Type 1 Diabetes; New-onset T1D; Newly Diagnosed Type 1 Diabetes Mellitus; Autoimmune diabetes; Thymoglobulin; ATG; Rabbit antithymocyte globulin
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Antilymphocyte Serum; thymoglobulin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antithymocyte globulin (Experimental): This group received a total of 6.5 mg/kg of antithymocyte globulin (e.g., Thymoglobulin®) divided into four doses as follows: Day 1, 0.5 mg/kg; Day 2, 2 mg/kg; Day 3, 2 mg/kg; and Day 4, 2 mg/kg.
  Interventions: Drug: Antithymocyte globulin
- Placebo (Placebo Comparator): This group received a saline solution to match the Thymoglobulin doses given to the active treatment group, on Day 1, 0.5 mg/kg; Day 2, 2 mg/kg; Day 3, 2 mg/kg; and Day 4, 2 mg/kg.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Antithymocyte globulin — Daily 4-day escalating dose
  Other Names: ATG; Thymoglobulin®; Rabbit antithymocyte globulin; RATG
  Arms: Antithymocyte globulin
Drug: Placebo — Daily 4-day saline solution
  Other Names: Inactive drug (pharmacologically); Saline solution
  Arms: Placebo

SUMMARY:
Antithymocyte globulin (e.g., Thymoglobulin®) is an antibody preparation that is commonly used to treat and prevent organ transplant rejection. The START trial aims to determine whether antithymocyte globulin (ATG) treatment can halt the progression of newly diagnosed type 1 diabetes when given within 12 weeks of disease diagnosis.

DETAILED DESCRIPTION:
Type 1 diabetes mellitus (T1DM) is an autoimmune disease in which the immune system mistakenly attacks the insulin-producing beta cells in the pancreas. Without these cells, the body cannot maintain proper blood glucose levels in response to daily activities, such as eating or exercise. Generally, at the time someone is diagnosed with T1DM, not all of a person's beta cells have been destroyed - between 15-40% remain healthy and are still able to produce insulin. Importantly, even small amounts of naturally produced insulin can improve blood sugar control, make daily management of diabetes less complicated, and reduce the risk of long term complications. Preserving the remaining precious beta cells is therefore the goal of the START trial.

The medication being tested in the START trial is antithymocyte globulin (e.g., Thymoglobulin®), a mixture of specialized proteins called antibodies. ATG attaches itself to white blood cells known as T cells, some of which are responsible for the immune system's attack on beta cells that occurs in T1DM. ATG can change how T cells work, and can eliminate a large proportion of the T cells from the bloodstream temporarily. Treatment of new onset T1DM with ATG is therefore expected to alter the behavior of the T cells to halt their attack, and also reduce T cell numbers, so that new T cells that grow in their place will learn to accept the beta cells, rather than attacking them.

Following an initial screening appointment, eligible participants will be randomly assigned to one of two groups: the Experimental Group will receive the study treatment while the Control Group that will receive placebo. Each participant has a 2 in 3 chance of being assigned to the treatment group, and a 1 in 3 chance of being assigned to the placebo. The START trial is a blinded study, so neither participants nor study physicians will know to which group an individual has been assigned. All participants will receive intensive diabetes management. Participants in both groups will be admitted to the hospital for 5-8 days to receive infusions of either the study drug or placebo.

The duration of the study is 2 years. Participants will have 8 follow-up appointments in the first year and 4 visits in the second year. Most of these visits will last 1- 2 hours. A review of interval health, a physical exam, an assessment of diabetes control including recent 5 day insulin use and blood sugar (e.g., glucose) testing, and blood collection for laboratory testing will occur at each visit. Four of the visits will last about 5 hours, during which participants will undergo mixed-meal tolerance testing (MMTT). This involves drinking a special drink, similar to a milkshake, and having blood specimens taken over a 4-hour period.

Subjects will be reimbursed for travel and parking expenses, and will receive compensation for their participation in the longer mixed meal tolerance test visits.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 diabetes (according to American Diabetes Association [ADA] criteria) within100 days of enrollment
* Positive for one or more autoantibodies (anti-glutamic acid decarboxylase [GAD], anti-insulin, or IA-2 autoantibodies)
* Peak stimulated C-peptide level >0.4 pmol/mL or >1.2ng/mL following an MMTT
* Serologic evidence of prior Epstein-Barr virus (EBV) infection (EBV seropositive)
* Willing to use acceptable forms of contraception

Exclusion Criteria:

* Any sign of active infection (e.g., hepatitis, tuberculosis, EBV, cytomegalovirus (CMV), or toxoplasmosis) at screening
* Positive for human immunodeficiency virus (HIV), tuberculosis, or hepatitis B surface antigen (HBsAg) at screening
* Prior history of any significant cardiac disease, such as congestive heart failure, arrhythmia, or structural defects, or suspicion thereof
* Use of glucocorticoids in the 28 days prior to study entry; or topical use of glucocorticoids
* Use of diabetes medications (other than insulin) that may affect glucose homeostasis, such as metformin, sulfonylureas, thiazolidinediones, or amylin
* Evidence of liver dysfunction
* Evidence of kidney disease
* Pregnancy or plan to become pregnant
* Leukopenia (<3,000 leukocytes/µL), neutropenia (<1,500neutrophils/µL), lymphopenia (<800 lymphocytes/µL), or thrombocytopenia (<125,000 platelets/µL).
* Prior treatment with rabbit ATG or known hypersensitivity or exposure to rabbit sera-derived products
* Vaccination with a live virus within the last 6 weeks before enrollment
* Prior or current therapy that is known to cause a significant, ongoing change in the course of T1DM or immunologic status
* Any condition that may compromise study participation or may confound the interpretation of the study results

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2007-08; Primary Completion 2012-06 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Gitelman, MD, Principal Investigator — University of California, San Francisco
Locations (9):
- United States (9):
  - Children's Hospital/USC School of Medicine, Los Angeles, California
  - Children's Hospital and Research Center, Oakland, California
  - UCSD/San Diego Children's Hospital, San Diego, California
  - Diabetes Center at UCSF, San Francisco, California
  - Barbara Davis Center for Childhood Diabetes, University of Colorado, Aurora, Colorado
  - Emory Children's Center, Atlanta, Georgia
  - University of Minnesota, Minneapolis, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - University of Pennsylvania/Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Participant level data and additional relevant materials are available to the public in TrialShare, the Immune Tolerance Network (ITN) Clinical Trials Research Portal. ITN TrialShare makes data from the consortium's clinical trials publicly available.

REFERENCES:
- [Background] Palmer JP, Fleming GA, Greenbaum CJ, Herold KC, Jansa LD, Kolb H, Lachin JM, Polonsky KS, Pozzilli P, Skyler JS, Steffes MW. C-peptide is the appropriate outcome measure for type 1 diabetes clinical trials to preserve beta-cell function: report of an ADA workshop, 21-22 October 2001. Diabetes. 2004 Jan;53(1):250-64. doi: 10.2337/diabetes.53.1.250. PMID 14693724
- [Background] Greenbaum CJ, Mandrup-Poulsen T, McGee PF, Battelino T, Haastert B, Ludvigsson J, Pozzilli P, Lachin JM, Kolb H; Type 1 Diabetes Trial Net Research Group; European C-Peptide Trial Study Group. Mixed-meal tolerance test versus glucagon stimulation test for the assessment of beta-cell function in therapeutic trials in type 1 diabetes. Diabetes Care. 2008 Oct;31(10):1966-71. doi: 10.2337/dc07-2451. Epub 2008 Jul 15. PMID 18628574
- [Result] Gitelman SE, Gottlieb PA, Rigby MR, Felner EI, Willi SM, Fisher LK, Moran A, Gottschalk M, Moore WV, Pinckney A, Keyes-Elstein L, Aggarwal S, Phippard D, Sayre PH, Ding L, Bluestone JA, Ehlers MR; START Study Team. Antithymocyte globulin treatment for patients with recent-onset type 1 diabetes: 12-month results of a randomised, placebo-controlled, phase 2 trial. Lancet Diabetes Endocrinol. 2013 Dec;1(4):306-16. doi: 10.1016/S2213-8587(13)70065-2. Epub 2013 Aug 28. PMID 24622416
- [Result] Gitelman SE, Gottlieb PA, Felner EI, Willi SM, Fisher LK, Moran A, Gottschalk M, Moore WV, Pinckney A, Keyes-Elstein L, Harris KM, Kanaparthi S, Phippard D, Ding L, Bluestone JA, Ehlers MR; ITN START Study Team. Antithymocyte globulin therapy for patients with recent-onset type 1 diabetes: 2 year results of a randomised trial. Diabetologia. 2016 Jun;59(6):1153-61. doi: 10.1007/s00125-016-3917-4. Epub 2016 Apr 6. PMID 27053235
- [Result] Salama A, Evanno G, Lim N, Rousse J, Le Berre L, Nicot A, Bach JM, Brouard S, Harris KM, Ehlers MR, Gitelman SE, Soulillou JP. Anti-Gal and Anti-Neu5Gc Responses in Nonimmunosuppressed Patients After Treatment With Rabbit Antithymocyte Polyclonal IgGs. Transplantation. 2017 Oct;101(10):2501-2507. doi: 10.1097/TP.0000000000001686. PMID 28198767
- [Derived] Boyle KD, Keyes-Elstein L, Ehlers MR, McNamara J, Rigby MR, Gitelman SE, Weiner LJ, Much KL, Herold KC. Two- and Four-Hour Tests Differ in Capture of C-Peptide Responses to a Mixed Meal in Type 1 Diabetes. Diabetes Care. 2016 Jun;39(6):e76-8. doi: 10.2337/dc15-2077. Epub 2016 Apr 13. No abstract available. PMID 27208317
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Click here for the Immune Tolerance Network (ITN) Web site — http://www.immunetolerance.org
- See also: ITN TrialShare: open public access to study level information — http://www.itntrialshare.org
- Available data/document: Individual Participant Data Set: START ITN028AI — http://www.itntrialshare.org/project/Studies/ITN028AIPUBLIC/Study%20Data/begin.view? — START ITN028AI is the Study Identifier in the Immune Tolerance Network (ITN) TrialShare Clinical Trials Research Portal
- Available data/document: Study Protocol: START ITN028AI — https://www.itntrialshare.org/project/Studies/ITN028AIPUBLIC/Study%20Data/begin.view?pageId=study.PARTICIPANTS — START ITN028AI is the Study Identifier in the Immune Tolerance Network (ITN) TrialShare Clinical Trials Research Portal
- Available data/document: Study overview, -data and reports, -manuscripts and abstracts, -availability of biospecimens, et al: START ITN028AI — https://www.itntrialshare.org/project/Studies/ITN028AIPUBLIC/Study%20Data/begin.view? — START ITN028AI is the Study Identifier in the Immune Tolerance Network (ITN) TrialShare Clinical Trials Research Portal

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited during an approximate 40-month accrual period. Initially 66 subjects were planned, however enrollment closed early at 58 subjects on June 30, 2011 secondary to slow accrual (planned 30-month accrual period).
Pre-assignment Details: Subjects ages 12 to 35 years who were first diagnosed with type 1 diabetes mellitus (T1DM) within 100 days of enrollment.
Groups:
- Antithymocyte Globulin: This group received a total of 6.5 mg/kg of antithymocyte globulin (Thymoglobulin®) administered intravenously and divided into four doses as follows: Day 1, 0.5 mg/kg; Day 2, 2 mg/kg; Day 3, 2 mg/kg; and Day 4, 2 mg/kg.
- Placebo: This group received a saline solution administered intravenously to match the antithymocyte globulin (Thymoglobulin®) doses given to the active treatment group, on Day 1, 0.5 mg/kg; Day 2, 2 mg/kg; Day 3, 2 mg/kg; and Day 4, 2 mg/kg.
Period: Overall Study
Arm/Group | Antithymocyte Globulin | Placebo
Started | 38 | 20
Completed | 35 | 16
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 0 | 4
Not completed — Withdrawal by Subject | 2 | 0
Not completed — IRB Recommendation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat
Groups:
- Total: Total of all reporting groups
Arm/Group | Antithymocyte Globulin | Placebo | Total
Number analyzed (Participants) | 38 | 20 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19 | 10 | 29
  Between 18 and 65 years | 19 | 10 | 29
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.4 (6.6) | 20.5 (7.1) | 19.8 (6.7)
Age, Customized [Number; unit: participants]
  12 -15 Years | 13 | 6 | 19
  16 - 21 Years | 13 | 6 | 19
  22 - 35 Years | 12 | 8 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 9 | 23
  Male | 24 | 11 | 35
Region of Enrollment [Number; unit: participants]
  United States | 38 | 20 | 58

OUTCOME MEASURES:

1. Primary Outcome: 2-Hour C-peptide Area Under the Curve (AUC) Result in Response to Standardized Mixed Meal Tolerance Test (MMTT)
Description: C-peptide is a substance released by the pancreas into the bloodstream in equal amounts to insulin and reflects how much insulin pancreatic beta cells are making. The standardized MMTT evaluates whether beta cells are producing endogenous insulin. The MMTT was performed in the morning and blood samples for C-peptide collected at baseline (pre-meal) and 15, 30, 60, 90, 120, 150, 180, 210,and 240 minutes post-meal. Results of the stimulated 2-hour (e.g., 120 minutes) post-meal C-peptide AUC are provided. Larger numbers are preferable (better) in these AUC results: more insulin being produced reflects less severe disease. C-peptide levels in the serum (e.g., AUC following a standardized MMTT) compared to control group at 1 year post treatment initiation for the evaluation of investigational products intended to preserve endogenous beta-cell function in T1DM trials is recognized by the Center for Drug Evaluation and Research (CDER) at the FDA as a valid efficacy primary endpoint.
Time Frame: Baseline (Pre-treatment initiation), Month 12
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: pmol/mL
Arm/Group | Antithymocyte Globulin | Placebo
Number analyzed (Participants) | 38 | 20
pmol/mL
  Baseline (Pre-treatment initiation) | 0.86 (0.37) | 0.93 (0.50)
  Month 12 | 0.66 (0.37) | 0.69 (0.52)
  Change from Baseline (Pre-treatment initiation) | -0.20 (0.29) | -0.24 (0.26)
Statistical Analysis 1: Comparison: Antithymocyte Globulin vs Placebo; Primary imputation method used for missing Month 12 AUC. Measuring range for C-peptide is 0.05-30 ng/mL; Test type: Superiority or Other; p = 0.60, ANCOVA — P-value is for testing treatment effect using an analysis of covariance with baseline ln(AUC+1) as a covariate and change in ln(AUC+1) from baseline as the outcome variable

2. Secondary Outcome: 4-Hour C-peptide Area Under the Curve (AUC) Result in Response to Standardized Mixed Meal Tolerance Test (MMTT)
Description: C-peptide is a substance released by the pancreas into the bloodstream in equal amounts to insulin and reflects how much insulin pancreatic beta cells are making. The standardized MMTT evaluates whether beta cells are producing endogenous insulin. The MMTT was performed in the morning and blood samples for C-peptide collected at baseline (pre-meal) and 15, 30, 60, 90, 120, 150, 180, 210,and 240 minutes post-meal. Results of the stimulated 4-hour (e.g., 240 minutes) post-meal C-peptide AUC are provided. Larger numbers are preferable (better) in these AUC results: more insulin being produced reflects less severe disease. C-peptide levels in the serum (e.g., AUC following a standardized MMTT) compared to control group at 1 year post treatment initiation for the evaluation of investigational products intended to preserve endogenous beta-cell function in T1DM trials is recognized by the Center for Drug Evaluation and Research (CDER) at the FDA as a valid efficacy endpoint.
Time Frame: Baseline (Pre-treatment initiation), Month 12
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: pmol/mL
Arm/Group | Antithymocyte Globulin | Placebo
Number analyzed (Participants) | 38 | 20
pmol/mL
  Baseline (Pre-treatment initiation) | 0.86 (0.30) | 0.90 (0.37)
  Month 12 | 0.67 (0.38) | 0.63 (0.39)
  Change from Baseline (Pre-treatment initiation) | -0.19 (0.30) | -0.27 (0.25)
Statistical Analysis 1: Comparison: Antithymocyte Globulin vs Placebo; Missing Month 12 AUC values were not imputed. Measuring range for C-peptide is 0.05-30 ng/mL; Test type: Superiority or Other; p = 0.40, ANCOVA — P-value is for testing treatment effect using an analysis of covariance with baseline In(AUC+1) as a covariate and change in In(AUC+1) from baseline as the outcome variable

3. Secondary Outcome: Insulin Use in Units Per Kilogram Body Weight Per Day
Description: The need to use exogenous insulin is an indication that the body is not producing enough endogenous insulin. Higher amounts of insulin use indicate higher disease activity.
Time Frame: Baseline (Pre-treatment), Months 12 and 24
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: units/day/kg
Arm/Group | Antithymocyte Globulin | Placebo
Number analyzed (Participants) | 38 | 20
units/day/kg
  Baseline (Pre-treatment initiation) | 0.34 (0.22) | 0.42 (0.24)
  Month 12 | 0.40 (0.24) | 0.49 (0.26)
  Change from Baseline to Month 12 | 0.07 (0.20) | 0.08 (0.20)
  Month 24 | 0.54 (0.31) | 0.47 (0.21)
  Change from Baseline to Month 24 | 0.19 (0.23) | 0.06 (0.25)
Statistical Analysis 1: Comparison: Antithymocyte Globulin vs Placebo; Comparison of groups for change from baseline (pre-treatment initiation) to Month 12; Test type: Superiority or Other; p = 0.59, ANCOVA — P-value is for testing treatment effect using an analysis of covariance with baseline level as a covariate and change in insulin use from baseline as the outcome variable
Statistical Analysis 2: Comparison: Antithymocyte Globulin vs Placebo; Comparison of groups for change from baseline (pre-treatment initiation) to Month 24; Test type: Superiority or Other; p = 0.14, ANCOVA — [p-value comment as in outcome 3, analysis 1]

4. Secondary Outcome: Number of Participants Who Are Exogenous-Insulin-Free
Description: as for outcome 3
Time Frame: Baseline (Pre-treatment), Months 12 , 18, and 24
Population: Intent-to-treat
Measure: Number; unit: participants
Arm/Group | Antithymocyte Globulin | Placebo
Number analyzed (Participants) | 38 | 20
participants
  Baseline (Pre-treatment initiation) | 1 | 0
  Month 12 | 1 | 0
  Month 18 | 1 | 0
  Month 24 | 1 | 0

5. Secondary Outcome: Number of Participants With Major Hypoglycemic Event(s) Post Treatment Randomization/Initiation
Description: Major hypoglycemic events are defined as a glucose concentration <55 mg/dL (grades 2-5, NCI-CTCAE version 3.0), or clinically: involving seizure(s) or involving loss of consciousness (coma), or requiring assistance from another individual in order to recover.
Time Frame: Baseline (Pre-treatment), Months 12 , and 24
Population: Intent-to-treat
Measure: Number; unit: participants
Arm/Group | Antithymocyte Globulin | Placebo
Number analyzed (Participants) | 38 | 20
participants
  Participants with Hypoglycemic Events Up to Mo. 12 | 23 | 12
  Participants with Hypoglycemic Events Up to Mo. 24 | 30 | 15
Statistical Analysis 1: Comparison: Antithymocyte Globulin vs Placebo; Comparison of groups up to Month 12; Test type: Superiority or Other; p > 0.099, Fisher Exact — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Antithymocyte Globulin vs Placebo; Comparison of groups up to Month 24; Test type: Superiority or Other; p = 0.75, Fisher Exact — [p-value comment as in outcome 3, analysis 1]

6. Secondary Outcome: 2-Hour and 4-Hour C-peptide Area Under the Curve (AUC) Results in Response to Standardized Mixed Meal Tolerance Test (MMTT)
Description: C-peptide is a substance released by the pancreas into the bloodstream in equal amounts to insulin and reflects how much insulin pancreatic beta cells are making. The standardized MMTT evaluates whether beta cells are producing endogenous insulin. The MMTT was performed in the morning and blood samples for C-peptide collected at baseline (pre-meal) and 15, 30, 60, 90, 120, 150, 180, 210,and 240 minutes post-meal. Results of the stimulated 2-hour (e.g., 120 minutes) and 4-hour (e.g., 240 minutes) post-meal C-peptide AUC are provided. Larger numbers are preferable (better) in these AUC results: more insulin being produced reflects less severe disease. C-peptide levels in the serum (e.g., AUC following a standardized MMTT) compared to control group at 1 year post treatment initiation for the evaluation of investigational products intended to preserve endogenous beta-cell function in T1DM trials is recognized by the CDER at the FDA as a valid efficacy endpoint.
Time Frame: Baseline (Pre-treatment), Month 24
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: pmol/mL
Arm/Group | Antithymocyte Globulin | Placebo
Number analyzed (Participants) | 38 | 20
pmol/mL
  Baseline (Pre-treatment initiation) | 0.86 (0.37) | 0.93 (0.50)
  2-hour AUC Month 24 | 0.58 (0.43) | 0.61 (0.67)
  Change from 2-hr MMTT Baseline | -0.27 (0.31) | -0.32 (0.32)
  4-hour AUC Month 24 | 0.56 (0.36) | 0.59 (0.63)
  Change from 4-hr MMTT Baseline | -0.26 (0.28) | -0.31 (0.38)
Statistical Analysis 1: Comparison: Antithymocyte Globulin vs Placebo; 2-Hour AUC change from baseline (pre-initiation treatment) to Month 24. Primary imputation method used for missing Month 24 AUC. Measuring range for C-peptide is 0.05-30 ng/mL; Test type: Superiority or Other; p = 0.38, ANCOVA — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Antithymocyte Globulin vs Placebo; 4-Hour AUC change from baseline (pre-initiation treatment) to Month 24. Missing Month 24 AUC values were not imputed. Measuring range for C-peptide is 0.05-30 ng/mL; Test type: Superiority or Other; p = 0.33, ANCOVA — [p-value comment as in outcome 2, analysis 1]

7. Secondary Outcome: Hemoglobin A1c
Description: Glycosylated hemoglobin (HbA1c) is a measure of the average plasma concentration of blood sugar (glucose) over the previous three months and measures the level of optimal management of underlying disease. An HbA1c of <=5.6% is considered normal. HbA1c of 6.5% or higher is typical for individuals with Type 1 Diabetes mellitus (T1DM).
Time Frame: Baseline (Pre-treatment), Months 12 and 24
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: Percentage (%)
Arm/Group | Antithymocyte Globulin | Placebo
Number analyzed (Participants) | 38 | 20
Percentage (%)
  Baseline (Pre-treatment initiation) | 6.7 (1.3) | 6.8 (1.2)
  Month 12 | 6.9 (1.6) | 7.7 (1.8)
  Change from Baseline to Month 12 | 0.1 (1.8) | 1.0 (1.5)
  Month 24 | 7.5 (1.5) | 8.2 (2.4)
  Change from Baseline to Month 24 | 0.6 (1.8) | 1.4 (1.9)
Statistical Analysis 1: Comparison: Antithymocyte Globulin vs Placebo; Comparison of groups for change from Baseline to Month 12; Test type: Superiority or Other; p = 0.07, ANCOVA — P-value is for testing treatment effect using an analysis of covariance with baseline level as a covariate and change in HbA1c from baseline as the outcome variable
Statistical Analysis 2: Comparison: Antithymocyte Globulin vs Placebo; Comparison of groups for change from Baseline to Month 24; Test type: Superiority or Other; p = 0.16, ANCOVA — [p-value comment as in outcome 7, analysis 1]

ADVERSE EVENTS:
Time Frame: From baseline (e.g., when informed consent signed) through study completion. The first participant enrolled in September 2007 and the last participant last visit for the study occurred in July 2013.
Description: Adverse Events (AEs) could be discovered through any of these methods:
  * Observing the participant.
  * Questioning the participant in an objective manner.
  * Receiving an unsolicited complaint from the participant.
Groups:
- Antithymocyte Globulin: This group received a total of 6.5 mg/kg of antithymocyte globulin (Thymoglobulin®) administered intravenously and divided into four doses as follows: Day 1, 0.5 mg/kg; Day 2, 2 mg/kg; Day 3, 2 mg/kg; and Day 4 2 mg/kg.
- Placebo: This group received a saline solution administered intravenously to match the antithymocyte globulin (Thymoglobulin®) doses given to the active treatment group, on Day 1, 0.5 mg/kg; Day 2, 2 mg/kg; Day 3, 2 mg/kg; and Day 4 2 mg/kg.
Arm/Group | Antithymocyte Globulin | Placebo
Serious Adverse Events (participants affected / at risk) | 9/38 | 4/20
Other Adverse Events (participants affected / at risk) | 38/38 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antithymocyte Globulin (N=38) | Placebo (N=20)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 0 (0)
Serum sickness (Immune system disorders) | 2 (2) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Salmonellosis (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Comminuted fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
CD4 lymphocytes decreased (Investigations) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (4) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Ketosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Affective disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (4) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1)
Mood altered (Psychiatric disorders) | 1 (1) | 0 (0)
Substance abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Axillary vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antithymocyte Globulin (N=38) | Placebo (N=20)
Leukopenia (Blood and lymphatic system disorders) | 14 (20) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 38 (48) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 9 (10) | 2 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (5) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Middle ear effusion (Ear and labyrinth disorders) | 0 (0) | 1 (2)
Eye irritation (Eye disorders) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 3 (3) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (6) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 3 (3)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (8) | 5 (7)
Oral disorder (Gastrointestinal disorders) | 2 (4) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (4) | 3 (3)
Catheter site pain (General disorders) | 5 (5) | 1 (1)
Chest discomfort (General disorders) | 3 (3) | 1 (1)
Chest pain (General disorders) | 2 (2) | 1 (1)
Face oedema (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (4) | 4 (5)
Influenza like illness (General disorders) | 2 (2) | 3 (3)
Infusion site pain (General disorders) | 1 (1) | 1 (1)
Infusion site swelling (General disorders) | 0 (0) | 1 (1)
Injection site discolouration (General disorders) | 0 (0) | 1 (1)
Injection site hypertrophy (General disorders) | 2 (2) | 0 (0)
Malaise (General disorders) | 2 (2) | 1 (1)
Pain (General disorders) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 6 (6) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 (3) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 36 (36) | 1 (1)
Seasonal allergy (Immune system disorders) | 7 (8) | 2 (2)
Serum sickness (Immune system disorders) | 36 (37) | 0 (0)
Bronchitis (Infections and infestations) | 4 (5) | 0 (0)
Ear infection (Infections and infestations) | 2 (2) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 1 (2)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1)
Gingival infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 3 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (5) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (2) | 2 (2)
Pharyngitis streptococcal (Infections and infestations) | 2 (3) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 5 (7) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 16 (32) | 7 (16)
Viral infection (Infections and infestations) | 5 (10) | 3 (3)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 4 (5) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint sprain (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 2 (3) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (4) | 0 (0)
CD4 lymphocytes decreased (Investigations) | 37 (37) | 0 (0)
Glycosylated haemoglobin increased (Investigations) | 0 (0) | 1 (1)
Haptoglobin increased (Investigations) | 2 (2) | 0 (0)
T-lymphocyte count decreased (Investigations) | 2 (2) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 7 (8) | 1 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 31 (493) | 16 (201)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 5 (6)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4) | 2 (2)
Dysaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 18 (25) | 10 (15)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 2 (3)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
Affective disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 3 (3) | 3 (3)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Restlessness (Psychiatric disorders) | 2 (2) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 2 (3) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 4 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 (13) | 5 (6)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 7 (8) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Lipoatrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (4)
Rash (Skin and subcutaneous tissue disorders) | 7 (8) | 2 (3)
Rash papular (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (5)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 3 (3)

LIMITATIONS AND CAVEATS:
Enrollment for this trial was closed at 58 participants and did not meet the planned sample size of 66 participants due to slow accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No